CLINICAL TRIAL: NCT06399523
Title: A Prospective, Randomized Controlled Clinical Trial to Evaluate the Efficacy of VR for Bipolar Disorder
Brief Title: A Study to Evaluate the Efficacy of VR for Bipolar Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Nanjing XR-Oasis Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YYLZ-CTP-001
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Bipolar Disorder; VR; Interventional Study
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR therapy (Experimental)
  Interventions: Device: VR therapy
- VR sham (Placebo Comparator)
  Interventions: Device: VR sham

INTERVENTIONS:
Device: VR therapy — Participants this group received additional VR therapy , with a total 20 sessions over a period of 4 weeks based on routine treatment.
  Arms: VR therapy
Device: VR sham — Participants in this group received additional VR sham(health education videos,a total of 20 health education videos over a period of 4 weeks) under virtual reality conditions on the basis of routine treatment.
  Arms: VR sham

SUMMARY:
Bipolar disorder is characterized by high morbidity, recurrence, disability, suicide and comorbidity rate which need novel, efficient, and safe treatment methods, and VR has demonstrate its efficacy in mental disease but not few focus on bipolar disorder. A prospective single center randomize clinical study therefore would be carried on to evaluate the efficacy of VR for Bipolar Disorder in China.

DETAILED DESCRIPTION:
Bipolar disorder (BD) refers to a type of mood disorder that clinically manifests as both manic or hypomanic episodes and depressive episodes. Bipolar disorder is characterized by high morbidity, recurrence, disability, suicide and comorbidity rate. The first episode often occurs before age 20, with a lifetime morbidity rate ranging from 1.5% to 6.4% . Patients with bipolar disorder spend significantly more time experiencing depressive episodes than manic or mixed symptoms throughout their lives. At the same time, depressive episodes can cause severe psycho-social disabilities, imposing a heavy economic burden on their families and society .

Despite being the first-line recommended treatment for bipolar depression, pharmacotherapy still cannot fully meet the clinical needs. Some patients do not achieve clinical remission even after receiving adequate and full-course pharmacotherapy. Even if clinical remission is achieved, many patients still have residual symptoms, and those in the maintenance phase still face a high risk of relapse. Psychotherapy has been reported to have various benefits such as improving interpersonal communication skills, enhancing cohesion, and building social support systems, and it has been widely used in the treatment of depression. Although psychological intervention plays a crucial role in the treatment of bipolar depression, its application in reality is still limited. One important reason is the shortage of psychological treatment service resources.

The application of virtual reality (VR) technology in the treatment of mental illnesses has overcome the limitations of traditional psychotherapy techniques. It provides a safer, more controllable, and personalized treatment approach, enabling patients to experience environments and events more intuitively and vividly. This study aims to explore the clinical intervention effects of a mental disorder adjuvant treatment software developed by Nanjing XR-Oasis Technology Co., Ltd. on patients with bipolar disorder experiencing depressive episodes. The technology is based on the theoretical frameworks of cognitive behavioral therapy, interpersonal therapy, mental health education, and Naikan therapy, combined with VR technology.

ELIGIBILITY:
Inclusion Criteria:

* 13 years or older
* Meet the diagnostic criteria for bipolar disorder - depressive episode in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* Able to understand the content of the scale
* Certain abilities in expressive, reading, and listening
* Total score of >17 on the Hamilton Rating Scale for Depression (HAMD-17)
* Inform consent

Exclusion Criteria:

* Poor physical condition unable to participate in the study
* Currently or previously diagnosed with other major mental disorders according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition（DSM-5）
* Severe or active physical illnesses that interfere with the study treatment
* Suicidal or self-harming ideas (defined as a score of >3 on item 3 of the Hamilton Depression Scale-17 suicide scale)
* Pregnant or lactating women
* Participate in other clinical trials within 1 month
* Epilepsy or severe eye diseases

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-04 (Estimated)

PRIMARY OUTCOMES:
Evolution of Depression | 1 month
  Changes in the total score of HAMD-17 at the end of the study compared to baseline

SECONDARY OUTCOMES:
Early Response | 2 weeks
  A reduction of ≥20% in the total score of HAMD-17 at the end of the 2nd week of treatment compared to baseline
Clinical Response | 2 months
  A reduction of ≥50% in the total score of HAMD-17 compared to baseline; specifically, sustained response is defined as a continuous reduction of ≥50% in the total score of HAMD-17 at the end of the 4th and 8th weeks of treatment compared to baseline
Clinical Remission | 2 months
  A total score of HAMD-17 ≤7; particularly, complete remission is defined as a total score of HAMD-17 ≤7 at the end of both the 4th and 8th weeks of treatment
Changes in the Clinical Global Impression Scale | 2 months
  Improvement (CGI-I) and Severity (CGI-S) scores compared to baseline
Conversion to mania | 2 months
  Change of A Young Mania Rating Scale(YMRS) >13 before and after treatment, and 1 month follow-up
Changes in Patient Satisfaction Scale | 2 months
  Changes in patients satisfaction scale before and after treatment, and 1 month follow-up
Change in biological rhythms | 2 months
  Change in Biological Rhythms Interview of Assessment in Neuropsychiatry(BRAIN) Scale before and after treatment, and 1 month follow-up
Change in Quality of life | 2 months
  Change in quality of life score before and after treatment, and 1 month follow-up
Intervention Acceptability | 2 months
  Acceptability was assessed by questions, "Rate the VR storyline on a scale of 0 to 5". Acceptability was measured with total score of the scale
Adverse Events | 2 months
  Change of Treatment Emergent Symptom Scale(TESS)before and after treatment, and 1 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The prescription data will not be shared with the public. However, if the intervention is effective, the educational materials will be released to the public.